CLINICAL TRIAL: NCT06394232
Title: A Phase 1/2a Multi-Center, Dose-Escalation Study to Evaluate the Safety & Efficacy of Eyecyte-RPE™ When Administered as a Single-dose Subretinal Injection in Subjects With Geographic Atrophy Secondary to Dry Age-related Macular Degeneration
Brief Title: Safety & Efficacy of Eyecyte-RPE™ in Patients With Geographic Atrophy Secondary to Dry Age-related Macular Degeneration.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eyestem Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ERPL-CTP-001
Record Dates: First submitted 2024-04-15; First posted 2024-05-01 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Retinal Disease; Macular Degeneration; Age-Related Macular Degeneration; Geographic Atrophy; Eye Diseases
Keywords: Age Related Macular Degeneration; Geographic Atrophy; Visual Impairment; Subretinal injection; Stem cells; Retinal Pigment Epithelial Cells
MeSH Terms: conditions — Retinal Diseases; Macular Degeneration; Geographic Atrophy; Eye Diseases; Vision Disorders | interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled into 3 sequential, ascending dose-level (DL) cohorts to enroll a maximum of 18 subjects.
  There will be three Cohorts
  1. DL1-Cohort 1: Eyecyte-RPE™ 100,000 cells
  2. DL2-Cohort 2: Eyecyte-RPE™ 200,000 cells
  3. DL3-Cohort 3: Eyecyte-RPE™ 300,000 cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 1-Cohort 1 (Experimental): Subjects who are allocated to Dose Level 1-Cohort 1 will receive 100,000 cells of Eyecyte-RPE™
  Interventions: Drug: Eyecyte-RPE™
- Dose Level 2-Cohort 2 (Experimental): Subjects who are allocated to Dose Level 2-Cohort 2 will receive 200,000 cells of Eyecyte-RPE™
  Interventions: Drug: Eyecyte-RPE™
- Dose Level 3-Cohort 3 (Experimental): Subjects who are allocated to Dose Level 3-Cohort 3 will receive 300,000 cells of Eyecyte-RPE™
  Interventions: Drug: Eyecyte-RPE™

INTERVENTIONS:
Drug: Eyecyte-RPE™ — Eyecyte-RPE™ is a suspension of hiPSCs (human induced Pluripotent Stem Cells) derived Retinal Pigment Epithelial Cells
  Other Names: Subretinal Injection; Oral Tacrolimus; Oral Mycophenolate Sodium

SUMMARY:
The goal of this clinical study is to evaluate the safety and efficacy of novel stem cell formulation in patients having Geographic Atrophy (GA) Secondary to Dry Age-related Macular Degeneration (d-AMD).

The main questions it aims to answer are:

* Safety and tolerability of the novel stem cell formulation
* Potential efficacy of the novel stem cell formulation

Participants will receive a single subretinal injection in their study eye and followed up for safety.

This is an India only study and the product is developed indigenously.

DETAILED DESCRIPTION:
Age-related Macular Degeneration (AMD) is a leading cause of vision impairment in the elderly and substantially affects the quality of life of an individual. Although the exact pathophysiological mechanisms behind the disease are multifactorial and complex, several genetic and environmental risk factors are associated with AMD, such as age, cigarette smoking, hypertension, abdominal obesity, dietary fat, and low physical activity.

Geographic Atrophy (GA) is the late stage of dry AMD(d-AMD). GA is a slow but inexorably progressive disease that causes irreversible blindness over time. Several new non-invasive tools such as Fundus Autofluorescence (FAF), Optical Coherence Tomography (OCT), and OCT Angiography (OCT-A) are being used to enable early diagnosis and follow up in these patients. Despite these advances, there are currently no approved treatments for GA that can replace the damaged RPE, photoreceptors, or outer retinal layers. In recent years, stem cell replacement therapy is being evaluated as an alternative to treat d-AMD.

In the pursuit to find a promising solution for d-AMD, which is an unmet medical need globally, Eyestem has been striving to develop a safe and effective stem-cell based therapy.

Theoretically, human induced pluripotent stem cells(hiPSCs) derived Eyecyte-RPE™, developed by Eyestem can help replace the damaged or lost retinal pigment epithelial (RPE) cells and potentially enable tissue regeneration in the diseased retina. In addition, stem cells can perform multiple functions, such as immunoregulation, prevention of apoptosis in sensory neurons, and secretion of neurotrophic factors. The latest stem cell transplantation studies performed by other research groups has been able to demonstrate that this therapy has a promising approach to restore visual function in eyes with degenerative retinal diseases.

The results of the pre-clinical safety and efficacy studies with Eyecyte-RPE™ have been very encouraging. It has been shown to provide significant beneficial effects on the degenerating retina in animals without any significant safety concerns, suggesting that this therapy may have substantial therapeutic value in d-AMD.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 50 years of age at Screening.
2. Diagnosis of Geographic Atrophy secondary to d-AMD
3. Have Best Corrected Visual Acuity (BCVA) equal to or less than 20/200 Snellen (ETDRS letter score ≤ 35) in the study eye at screening.

   1. Phase 1 ≤ 20/200 and
   2. Phase 2a ≥ 20/64 (ETDRS letter score 60) in the study eye at Screening.
4. Vision in the unoperated eye must be better or equal to vision in the study eye.
5. Willing, committed, and able to return for ALL clinic visits and complete all study related procedures.
6. Be medically suitable to undergo anesthesia, vitrectomy and subretinal injection in the opinion of the Investigator.
7. Be medically suitable for immunosuppression therapy in accordance with the requirements of this protocol in the opinion of the Investigator.
8. Able to read (or if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member) and understand, and willing to sign the informed consent form (ICF)
9. Willing to provide signed Informed Consent prior to any procedures being performed at Visit 1, Screening.
10. Negative for HIV, HbsAg, HCV, TB
11. The GA lesion must meet the following criteria as determined by the central reading center's assessment of Fundus Autofluorescence (FAF) imaging at screening:

    1. Total GA area must be ≥ 1.25 and ≤ 17.5 mm2 (0.5 and 7 disk areas [DA] respectively)
    2. The entire GA lesion must be completely visualized on the macula centered image and must be able to be imaged in its entirety and not contiguous with any areas of peripapillary atrophy.
    3. At least one of the lesions has to be sub-foveal.

Exclusion Criteria:

1. Have evidence of neovascular AMD in either eye by clinical examination, fluorescein angiography or optical coherence tomography.
2. Have GA secondary to a condition other than AMD such as Stargardt disease, cone rod dystrophy or toxic maculopathies like Chloroquine maculopathy in either eye.
3. Have any evidence of active or inactive choroidal neovascularization (CNV) due to other causes such as ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, uveitis, punctate inner choroidopathy, or multifocal choroiditis in the study eye.
4. Axial myopia greater than -6 diopters or axial length more than 26 mm.
5. Have a decrease in BCVA in the study eye due to causes other than GA (e.g., pigment abnormalities, dense sub foveal hard exudates, previous vitreoretinal surgery, retinal dystrophies, non-retinal conditions, visually significant cataract, macular ischemia, etc.).
6. Have the presence of retinal pigment epithelial tears or rips involving the macula in the study eye at screening.
7. Have a history or evidence of vitreous hemorrhage in the study eye.
8. Have a history or clinical evidence of severe diabetic retinopathy, diabetic macular edema, retinal vein occlusion or any other vascular disease affecting the retina in the study eye.
9. Have had a prior pars plana vitrectomy in the study eye.
10. Have a history of retinal detachment or treatment or surgery for retinal detachment in the study eye.
11. Have history of a macular hole in the study eye.
12. Have had any other ocular surgery (except cataract) within 2 months or Yttrium Aluminum Garnet (YAG) laser capsulotomy in the study eye in the past 4 weeks.
13. Have had a prior trabeculectomy or other filtration surgery in the study eye.
14. History of any form of glaucoma in the study eye.
15. Patients with ocular pathology, particularly that of retina (other than AMD).
16. Have active intraocular inflammation or a history or evidence of uveitis in either eye.
17. Have active ocular or periocular infection in either eye, or a history of any ocular or periocular infection within the 2 weeks prior to Visit 1, Screening in either eye.
18. Have a history of scleromalacia in either eye.
19. Have had previous therapeutic radiation in the study eye.
20. Have a history of corneal transplant or corneal dystrophy.
21. Have any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the subject beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
22. Have a history of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications.
23. Have participated as a subject in any clinical study within 6 months prior to Day 0, Baseline.
24. Have a known serious allergy to fluorescein sodium for injection in angiography, Povidone Iodine or any of the other medications required for anesthesia or the subretinal injection procedure.
25. Be a female who is pregnant, breastfeeding, or of childbearing potential, unwilling to practice adequate contraception throughout the study at Screening and Baseline.
26. Currently receiving aspirin, aspirin containing products and/or any other coagulation modifying drugs which cannot be discontinued 7 days prior to surgery.
27. Have any systemic condition that would qualify the subject as being immunocompromised (e.g., severely uncontrolled diabetes, cancer).
28. Patients with Optic Atrophy

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Fundus Autofluorescence- | Upto 12 months
  Overall change in the geographic atrophy (GA) lesion area of the study eye over time using Fundus Autofluorescence (FAF)

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA)-Mean change from baseline in BCVA score in study eye and fellow eye. | Upto 12 months
  Change from baseline over time in BCVA as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The BCVA score (in letter units) will be reported.
Spectral-Domain Optical Coherence Tomography (SD-OCT)-Mean change from baseline in the Geographic Atrophy (GA) area in study eye and fellow eye | Upto 12 months
  Overall change in the GA lesion area of the study eye over time using SD-OCT
Fundus Photography- Changes between study eye and fellow eye | Upto 12 months
  Correlation assessment between quantitative metrics derived from Color fundus photography images
Microperimetry-Mean change from baseline in mean sensitivity | Upto 12 months
  Change from initial assessment over time in retinal sensitivity, as assessed by Microperimetry (MP)
National Eye Institute-Visual Function Questionnaire Quality of Life score | Upto 12 months
  Change over time in National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) Quality of Life (QoL) score

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Shri Ganapati Netralaya, Jālna, Maharashtra
  - All India Institute of Medical Sciences, Delhi, New Delhi
  - L V Prasad Eye Institute, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soundararajan L, Surendran H, Patlolla N, Battu R, Stoddard J, Arrizabalaga S, Liu Z, Lingam G, Su X, Ryals RC, Pal R. Allogeneic RPE cell suspension manufactured at scale demonstrating preclinical safety and efficacy led to IND approval. NPJ Regen Med. 2025 Apr 19;10(1):19. doi: 10.1038/s41536-025-00407-0. PMID 40253438